CLINICAL TRIAL: NCT06577194
Title: A Single-Center, Single-Arm Study of Neoadjuvant Short-Course Radiotherapy With IL-2 Followed by Sequential Immunotherapy With CAPOX Combined With PD-1 Antibody and IL-2 for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRSYM20240827
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-01

CONDITIONS: Rectal Cancer; Advanced Solid Tumor
Keywords: Immunotherapy; Short-course radiotherapy; IL-2
MeSH Terms: conditions — Rectal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Experimental arm
  Interventions: Drug: Sintilimab + IL-2 Combined with CAPOX; Radiation: Short-course radiotherapy

INTERVENTIONS:
Drug: Sintilimab + IL-2 Combined with CAPOX — Sintilimab + IL-2 Combined with Capox
Radiation: Short-course radiotherapy — Short-course radiotherapy+IL-2

SUMMARY:
A Single-Center, Single-Arm Study of Neoadjuvant Short-Course Radiotherapy with IL-2 Followed by Sequential Immunotherapy with CAPOX Combined with PD-1 antibody and IL-2 for Locally Advanced Rectal Cancer

DETAILED DESCRIPTION:
Globally, there are around 732,000 new cases of rectal cancer annually, with locally advanced rectal cancer (T3-4 or N+) comprising a significant proportion. The current NCCN guidelines recommend neoadjuvant chemoradiotherapy followed by total mesorectal excision (TME) and adjuvant chemotherapy, which has significantly reduced local recurrence rates from over 30% to less than 10%. However, challenges such as low rates of functional sphincter preservation, high incidence of distant metastasis, and limited long-term survival benefits persist. In response, total neoadjuvant therapy (TNT)-completing all chemotherapy and radiotherapy before surgery-has emerged as a strategy to improve outcomes. Yet, TNT may not be suitable for all patients due to the risk of overtreatment and associated toxicities.

Immunotherapy, including adoptive cell transfer (ACT) and immune checkpoint blockade (ICB), offers new therapeutic avenues for locally advanced rectal cancer. However, most colorectal cancer patients show limited responses to immunotherapy. For example, ACT has shown suboptimal results due to poor T-cell infiltration in tumors, and only a small subset of patients benefit from immune checkpoint inhibitors (ICIs). While PD-1/PD-L1 inhibitors are effective in mismatch repair-deficient (dMMR) or microsatellite instability-high (MSI-H) colorectal cancer, MSI-H tumors account for less than 5% of rectal cancer cases. Consequently, most patients with microsatellite-stable (MSS) tumors gain minimal benefit from monotherapy.

Immunotherapy resistance in MSS colorectal cancer is attributed to low tumor mutational burden, poor T-cell infiltration, and an immunosuppressive tumor microenvironment (iTME). Strategies to enhance local immune cell infiltration and reverse the iTME are crucial for improving immunotherapy efficacy in these cases. For instance, radiotherapy can synergize with immunotherapy by releasing tumor antigens and reshaping the immune environment to boost antitumor responses. Studies like UNION and TORCH have shown promising results by combining neoadjuvant chemoradiotherapy with anti-PD-1 immunotherapy in pMMR/MSS locally advanced rectal cancer patients.

Interleukin-2 (IL-2) plays a critical role in immune regulation, promoting T-cell growth and differentiation and enhancing cytotoxic T lymphocyte (CTL) and natural killer (NK) cell activity. High-dose IL-2 therapy has been used to treat malignant melanoma and renal cell carcinoma, leading to long-term survival in about 15% of patients. However, this approach is limited by severe side effects, such as hypotension and capillary leak syndrome. Current research focuses on improving IL-2 efficacy at low doses, including developing IL-2 variants with enhanced selectivity to avoid regulatory T cell (Treg) activation. Additionally, combining IL-2 with other treatments has shown significant clinical benefits. For example, in chronic lymphocytic choriomeningitis virus infection (LCMV), PD-1 and IL-2 combination therapy demonstrated superior efficacy compared to monotherapy. Preclinical studies in tumors also showed that PD-1/IL-2 combination therapy reversed terminal T-cell exhaustion, generating effector CD8+ T cells with enhanced profiles.

Based on these findings, combining IL-2 with anti-PD-1 therapy provides a strong foundation for clinical trials in locally advanced rectal cancer, specifically using neoadjuvant short-course radiotherapy combined with IL-2, followed by CAPOX, PD-1 monoclonal antibodies, and IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 70 years;
* ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1;
* Tumor tissue samples obtained and histologically confirmed as rectal adenocarcinoma;
* Adequate hematological, liver, and kidney functions: neutrophil count ≥ 1.5×10^9/L; platelet count ≥ 75×10^9/L; serum total bilirubin ≤ 1.5× upper limit of normal (UNL); aspartate aminotransferase ≤ 2.5× UNL; alanine aminotransferase ≤ 2.5× UNL; serum creatinine ≤ 1.5× UNL.

Exclusion Criteria:

* Metastatic disease (Stage IV);
* Recurrent rectal cancer;
* Concurrent active bleeding, perforation, or other complex situations that cannot be addressed with emergency colostomy surgery alone;
* Previous systemic anti-cancer treatment for colorectal cancer;
* Coexistence of other non-colorectal cancer malignancies;
* Patients with any active autoimmune diseases, or a history of needing steroids or immunosuppressive drugs;
* Patients with interstitial lung disease, non-infectious pneumonia, or uncontrolled systemic diseases (e.g., diabetes, hypertension, pulmonary fibrosis, and acute pneumonia);
* Previous treatment-induced any grade 2 or above toxicity reaction (according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5 classification) that has not subsided (excluding anemia, hair loss, and skin pigmentation);
* Previous treatment with anti-programmed death receptor-1 (PD-1) or its ligand (PD-L1) antibodies, anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) antibodies;
* Pregnant or breastfeeding women;
* Known or tested positive for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Known or suspected allergy history to any drugs used in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission | Two years
  The rate of pathological complete remission (pCR) plus clinical complete remission (cCR).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No